CLINICAL TRIAL: NCT01122914
Title: A Pilot Study Using Anakinra/Kineret for the Treatment of Patients With Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100100; 10-I-0100
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-04-07

CONDITIONS: Anakinra; Kineret; Atopic Dermatitis; Eczema; Allergic Disease
Keywords: Kineret; Anakinra; Atopic Dermatitis; Eczema; Allergic Disease
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Interleukin 1 Receptor Antagonist Protein

INTERVENTIONS:
Drug: Anakinra

SUMMARY:
Background:

* Severe atopic dermatitis, also known as eczema, is a chronic inflammatory skin condition that affects both children and adults and causes severe itching and skin redness. Current treatments of atopic dermatitis include topical creams and lotions, light therapy, and medications. However, the difficulty with long-term treatment for the chronic and severe nature of the disease requires more effective and better-tolerated therapeutic options.
* Anakinra is a drug that blocks a substance called interleukin-1 (IL-1), which may be important in causing the inflammation in atopic dermatitis. Researchers are interested in determining whether anakinra can be used to help treat atopic dermatitis. Anakinra has been approved by the Food and Drug Administration to treat rheumatoid arthritis in adults and children, but it has not been approved for use in adults or children with atopic dermatitis and is considered an experimental treatment in this study. In this study Anakinra will be administered as an injection under the skin every day for 3 months

Objectives:

- To assess the safety and effectiveness of using anakinra to treat severe atopic dermatitis in children.

Eligibility:

- Children between 10 and 18 years of age who have been diagnosed with severe atopic dermatitis that has not responded to standard treatment.

Design:

* Initial Screening: Participants will have an initial screening visit with a complete physical examination and medical history, blood and urine tests, photographs of the skin ,skin biopsy, and other tests as required.
* Run-in Period: At the screening visit, participants will receive a diary card and will be asked to track their atopic dermatitis symptoms on standard treatment for 2 months.
* Start of Treatment: At the end of the 2 month Run-in period participants will return for an inpatient visit (2 days) to receive the initial dose of anakinra and will be watched for any side effects. During the inpatient visit, participants will have additional examinations and blood and urine tests, and will be instructed on how to administer the anakinra injections at home.

Treatment Period: - Participants will return once a week for the first 2 weeks of treatment, at the end of the first month, and then once a month for the following 2 months, for a physical exam and blood tests. Participants will be asked to record symptoms related to their atopic dermatitis, anakinra administration and any side effects related to the anakinra on the diary card. The diary cards will be reviewed and collected at each visit.-

End of Treatment Period: At the end of 3 months of treatment with anakinra, participants will again be asked to record symptoms related to their atopic dermatitis on the diary card. Participants will be seen once a month for 3 months for a physical exam, blood tests and review of the diary card. . The final study visit will take place at the end of the 3rd month and will include a physical exam, blood tests, photographs and skin biopsy.

DETAILED DESCRIPTION:
Severe refractory atopic dermatitis is a chronic inflammatory pruritic skin condition that affects both children and adults. The disease is marked by periods of exacerbation and remission. Symptoms of atopic dermatitis may resolve by adolescence; however, it is estimated that the disease may persist in 50 percent of affected children well into adulthood.

Current possible treatments of atopic dermatitis include the use of topical corticosteroids, calcineurin inhibitors, phototherapy, as well as systemic medications i.e., methotrexate, cyclosporine, azathioprine, mycophenolate mofetil and interferon gamma. The difficulty with long-term treatment of this disease lies in its chronic nature associated with severe episodes. The combination of chronicity and severity of episodes of this diseases demands more effective and better-tolerated therapeutic options than those that are currently available. While the pathways of allergic inflammation are different than those of other inflammatory conditions, certain elements may overlap, providing targets for immune modulation. One of these targets is the interleukin-1 (IL-1) receptor.

The IL-1 receptor plays an important role in the development and maintenance of Th2 responses. Genetic, in vivo and in vitro data demonstrate a significant role for IL-1 signaling allergic and skin inflammatory conditions. This pilot study is therefore designed to assess the safety and efficacy of IL-1ra, a natural inhibitor of the IL-1 receptor, in disrupting atopic pathophysiologic pathways. Specifically, we will treat severe refractory atopic dermatitis associated with evidence of multiple specific allergic sensitivities. Up to 8 patients ages 10-30 with severe refractory dermatitis will be enrolled. Patients will be initially evaluated to establish the diagnosis of severe refractory AD as evidenced by SCORAD score greater than 40, followed by a 2 month (8 week) run-in period, a 3 month (12 week) treatment period of 3mg/kg/day anakinra given subcutaneously, followed by a 3 month (12 week) post-treatment evaluation period. In order to be considered evaluable for response, patients must have received a minimum of 67 out of 84 doses (80 percent) of anakinra. The primary endpoint is lack of an increase in serious infections, the secondary endpoint is a reduction of 30 percent or more in SCORAD score, and tertiary endpoints are cellular phenotypic and cytokine responses to IL-1 receptor blockade in atopic patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for enrollment in this protocol, participants must fulfill all of the following criteria:

1. Must be 10 years to 30 years of age
2. Patient or legal guardian must be able to give informed consent
3. Must have evidence of severe atopic dermatitis as determined by the investigators and a SCORAD score >40 performed within 90 days of study entry
4. Must have report from primary physician documenting lack of sufficient response to topical corticosteroids for > 6 months
5. Must have skin test or radioallergosorbent test (RAST) showing sensitivity to greater than or equal to 3 food and/or airborne allergens
6. Must have a baseline CBC that demonstrates:

   * White Blood Cell Count (WBC) greater than or equal to lower limit of normal for age
   * Absolute Neutrophil Count (ANC) greater than or equal to lower limit of normal for age

     c. Platelet Count greater than or equal to lower limit of normal for age
7. Must not be pregnant or breastfeeding
8. If subject is a female that has begun menstruation, and is sexually active, she must agree to consistently use contraception throughout study participation. Acceptable forms of contraception are:

   * Condoms, male or female, with spermicide
   * Diaphragm or cervical cap with spermicide
   * Intrauterine device
   * Contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method
   * Male partner has previously undergone a vasectomy for which there is documentation of aspermatogenic sterility
   * Abstinence
9. Must have a primary care physician
10. Must be willing to submit blood and skin tissue for storage

EXCLUSION CRITERIA:

A patient will be ineligible to participate in this protocol if any of the following criteria are fulfilled:

1. Patient is taking oral or injectable immunomodulators (such as methotrexate, imuran, and cyclosporine) or biologics (such as etanercept or omalizumab).
2. Patient requires systemic immunosuppression at any time during the study
3. Patient has known diseases of immunodysregulation or immunodeficiency.
4. Any chronic medical condition other than atopic dermatitis, allergy/asthma and infection, such as heart disease, diabetes and autoimmunity that, in the investigator s opinion, places the patient at undue risk by participating in the study.
5. History of anaphylactic reaction or hypersensitivity to anakinra.
6. The presence of certain types of acquired abnormalities of immunity such as human immunodeficiency virus (HIV), cytotoxic chemotherapy for malignancy could be grounds for possible exclusion if, in the opinion of the investigator, the presence of such disease process interferes with evaluating a coexisting abnormality of immunity that is a subject of study under this protocol.
7. The presence of any dermatologic diagnosis which, in the investigator's opinion, is not consistent with atopic dermatitis and would impair the ability to assess drug response.
8. Has a diagnosis of active tuberculosis with consistent findings from a PPD skin test, computerized tomography (CT) scan or Chest x-ray. Those subjects found to have a positive PPD will be referred back to their primary care physician for appropriate management.
9. Has received a live vaccine within 4 weeks prior to therapy or potential need for a live vaccine during the study.
10. Is unwilling to undergo testing or procedures associated with this protocol.
11. The patient or guardian is unable or unwilling to give daily injections.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2010-04-14; Primary Completion 2015-04-07 (Actual); Study Completion 2015-04-07 (Actual)

PRIMARY OUTCOMES:
Improvement of Atopic Dermatitis symptoms without increase in serious infections; Response to treatment with a 30 percent decrease in SCORAD score. | 2 years

SECONDARY OUTCOMES:
Determine immunological phenotype and cytokine profile of peripheral blood before and after treatment with Anakinra; Determine impact of IL-1 r neutralization on total and antigen specific allergen sensitivity. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Milner, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Leung DY, Boguniewicz M, Howell MD, Nomura I, Hamid QA. New insights into atopic dermatitis. J Clin Invest. 2004 Mar;113(5):651-7. doi: 10.1172/JCI21060. PMID 14991059
- [Background] Adjers K, Pessi T, Karjalainen J, Huhtala H, Hurme M. Epistatic effect of IL1A and IL4RA genes on the risk of atopy. J Allergy Clin Immunol. 2004 Mar;113(3):445-7. doi: 10.1016/j.jaci.2003.12.582. PMID 15007345
- [Background] Schmitt J, Schakel K, Schmitt N, Meurer M. Systemic treatment of severe atopic eczema: a systematic review. Acta Derm Venereol. 2007;87(2):100-11. doi: 10.2340/00015555-0207. PMID 17340015